CLINICAL TRIAL: NCT03860961
Title: Increasing the Dose of Survivorship Care Planning in Prostate Cancer Survivors Who Receive Androgen Deprivation Therapy
Brief Title: Increasing the Dose of Survivorship Care Planning in Improving Care and Outcomes in Prostate Cancer Survivors Receiving Androgen Deprivation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NRG-CC007CD; NCI-2019-00794 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-CC007CD (Other: NRG Oncology); NRG-CC007CD (Other: DCP); NRG-CC007CD (Other: CTEP); UG1CA189867 (NIH)
Record Dates: First submitted 2019-02-26; First posted 2019-03-04 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-09

CONDITIONS: Prostate Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Survivorship Care Plan) (Active Comparator): Practices review a Survivorship Care Plan (SCP) with patients and send it to the primary care physician (PCP) during the last week of radiation therapy (RT).
  Interventions: Other: Survivorship Care Plan
- Arm B (Enhanced Survivorship Care Plan) (Experimental): Practices review a treatment plan (TP) with patients and send it to the PCP at the beginning of RT. Practices also review a SCP as in arm A.
  Interventions: Other: Survivorship Care Plan; Other: Treatment Plan

INTERVENTIONS:
Other: Survivorship Care Plan — Given survivorship care plan
Other: Treatment Plan — Given treatment plan
  Arms: Arm B (Enhanced Survivorship Care Plan)

SUMMARY:
This trial studies how well increasing the dose of survivorship care planning improves care and outcomes in prostate cancer survivors receiving radiation therapy and androgen deprivation therapy. There is a need for coordinated care between the cancer care team with the primary care team. This is especially important for prostate cancer survivors who need routine cancer care follow-up with their radiation oncologist and also coordinated routine follow-up with their primary care provider (PCP). This is important because androgen deprivation therapy increases a patient's risk for developing diabetes, hypercholesterolemia, and cardiovascular events. Increasing the dose of survivorship may improve care and outcomes of cancer survivors than standard practices.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the experimental arm (increased doses of survivorship care planning [SCP]) has more patients who saw a primary care provider and had blood glucose and cholesterol checked in year 2 (13-24 months) after finishing radiation therapy (RT) as compared to the control arm.

SECONDARY OBJECTIVES:

I. To determine if patients who receive increased doses of SCP have lower cardiovascular disease (CVD) risk score at 2 years as compared to patients who receive a one-time SCP.

II. To determine if patients who receive increased doses of SCP have improved patient reported coordination and satisfaction with care with respect to their primary care provider (PCP) or cardiologist as compared to patients who receive a one-time SCP and whether health literacy modifies the effect of SCP use on patient-reported coordination of care and satisfaction with care with respect to their PCP or cardiologist.

III. To determine the number of patients eligible, but without a PCP/cardiologist.

IV. To describe the current practice related to SCP delivery and prostate cancer survivor monitoring in participating National Cancer Institute (NCI) Community Oncology Research Program (NCORP) practices.

EXPLORATORY OBJECTIVE:

I. To determine if patients who receive increased doses of SCP have improved patient reported coordination and satisfaction with care with respect to their cancer specialist as compared to patients who receive a one-time SCP and whether health literacy modifies the effect of SCP use on patient-reported coordination of care and satisfaction with care with respect to their cancer specialist.

Practices are randomized to 1 of 2 arms. After completion of study, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* PRACTICE ELIGIBILITY CRITERIA
* All institutions participating in a practice are NCORP components or sub-components
* Have a mechanism for delivering SCPs to prostate cancer patients. Practices that currently provide SCPs are eligible but for this trial will need to use the study-provided SCP template.
* See at least 10 patients meeting eligibility criteria per year.
* Completion and submission of the NRG-CC007CD Letter of Intent (LOI) (posted on the Cancer Trials Support Unit [CTSU] website) by each practice to NRGCC007CD@nrgoncology.org).
* Institutional Review Board (IRB) approval
* Each principal investigator (PI) and research assistant (RA) at a NCORP practice must complete NRG-CC007CD SCP training. A training certificate will need to be completed and uploaded to the CTSU Regulatory Submission Portal. (See NRG-CC007CD Training Memo and Slides; located on the CTSU website). Note: staff and physicians cannot be part of multiple practices
* For a practice that is participating on Wake Forest study, WF-1804CD is not able to participate in this trial in order to not impact the fidelity of either trial. As long as the clinicians (physicians, American Physician Partners [APPs]) are different for the patient populations of the two trials, a practice is eligible to participate in both trials
* PATIENT ELIGIBILITY CRITERIA - PRIOR TO REGISTRATION (STEP 1)
* The participant must be able to complete required questionnaires in English
* The participant must have a diagnosis of prostate adenocarcinoma that will be treated with RT plus androgen deprivation therapy (ADT) with curative intent. Both definitive RT (intact prostate) and postprostatectomy RT patients are eligible

  * The ADT must be planned for at least 4 months and must include luteinizing hormone-releasing hormone (LHRH) agonist or LHRH antagonist
  * ADT may have started for no more than 120 days before registration
* The participant must have a primary care provider and/or cardiologist or plan to obtain one
* Comorbidities assessed at study entry using the Adult Comorbidity Evaluation (ACE)-27 instrument (located on the CTSU website)
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2025-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald C Chen, Principal Investigator — NRG Oncology
Locations (79):
- United States (79):
  - Kingman Regional Medical Center, Kingman, Arizona
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Augusta University Medical Center, Augusta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Hunterdon Medical Center, Flemington, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Novant Cancer Institute Radiation Oncology - Supply, Supply, North Carolina
  - Novant Health Cancer Institute Radiation Oncology - Wilmington, Wilmington, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 833 participants screened at randomized practices, 550 were enrolled.
Units Other Than Participants: Practices
Period: Overall Study
Arm/Group | Arm A (Survivorship Care Plan) | Arm B (Enhanced Survivorship Care Plan)
Started | 277; 18 Practices | 273; 17 Practices
Completed (Number of participants evaluable for the primary endpoint) | 257; 18 Practices | 256; 17 Practices
Not Completed | 20; 0 Practices | 17; 0 Practices
Not completed — Withdrawal by Subject | 6 | 11
Not completed — Death | 10 | 6
Not completed — Incomplete two-year data | 4 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled participants
Groups:
- Arm A (SCP): Practices review a SCP with patients and send it to the PCP during the last week of RT.
- Arm B (Enhanced SCP): Practices review a treatment plan (TP) with patients and send it to the PCP at the beginning of RT. Practices also review a SCP as in arm A.
- Total: Total of all reporting groups
Arm/Group | Arm A (SCP) | Arm B (Enhanced SCP) | Total
Number analyzed (Participants) | 277 | 273 | 550
Age, Continuous [Mean (Full Range); unit: years] | 70 [49 to 88] | 70 [53 to 91] | 70 [49 to 91]
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 70 | 61 | 131
  ≥ 65 years | 207 | 212 | 419
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 277 | 273 | 550
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 9
  Not Hispanic or Latino | 268 | 261 | 529
  Unknown or Not Reported | 7 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39 | 42 | 81
  White | 229 | 220 | 449
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 6 | 5 | 11
Past smoker [Count of Participants; unit: Participants] | 142 | 139 | 281
Current smoker [Count of Participants; unit: Participants] | 31 | 33 | 64
Uses hypertension medication [Count of Participants; unit: Participants] | 187 | 179 | 366
Has Diabetes [Count of Participants; unit: Participants] | 70 | 72 | 142
Number of comorbidities determined by the Adult Comorbitity Evaluation-27 (ACE-27) [Count of Participants; unit: Participants] — The Adult Comorbidity Evaluation-27 (ACE-27) is a tool used to assess comorbid conditions in adult patients, particularly in the context of cancer care. For this study it is utilized here only to determine the number of comorbid conditions rather to than to calculate a score based on both the presence and severity of such conditions.
  Participants
    ≤ 2 | 185 | 181 | 366
    >2 | 92 | 92 | 184
Health Literacy Level determined by Brief Health Literacy Screen (BHLS) [Count of Participants; unit: Participants] — BHLS is a validated instrument that consists of three questions on a 5-point response scale. The total score ranges from 3 to 15, by which participants are then categorized as having inadequate, marginal, or adequate health literacy. Population: Due to incomplete questionnaires, the BHLS score was not able to be calculated for all participants.
  Participants
    number analyzed (Participants) | 276 | 271 | 547
    Inadequate | 30 | 35 | 65
    Marginal | 45 | 61 | 106
    Adequate | 201 | 175 | 376

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Adhering to Cardiovascular Follow-up Recommendations in the Second Year After Radiation Treatment
Description: A joint publication from the American Heart Association, American Cancer Society and American Urological Association made specific recommendations regarding cardiovascular follow-up for prostate cancer patients who receive androgen deprivation therapy (ADT) (Levine, 2010). Medical records from each participant's primary care physician (PCP) and cardiologist were reviewed to determine if a participant received care that followed the guideline recommendations interpreted in this study as meeting all three of the following criteria:
  * saw a primary care provider (PCP) or cardiologist
  * had fasting blood glucose checked
  * had fasting cholesterol check.
Time Frame: During the second year (13 to 24 months) after completion of approximately 4-9 weeks of radiation therapy.
Population: Eligible participants from randomized practices with necessary data for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A (Survivorship Care Plan): Practices review a SCP with patients and send it to the PCP during the last week of RT.
Arm/Group | Arm A (Survivorship Care Plan) | Arm B (Enhanced Survivorship Care Plan)
Number analyzed (Participants) | 257 | 256
Participants | 160 | 157
Statistical Analysis 1: Comparison: Arm A (Survivorship Care Plan) vs Arm B (Enhanced Survivorship Care Plan); Cluster-randomized trial, cluster=practice, maximum 25 patients/practice. Assuming 14 pts/practice, cluster size coefficient of variation of 0.5, intra-cluster correlation (ρ) of 0.04, design effect 1.51, and 59.8% of Arm A patients meeting the criteria provides 80% power for a two-sided α=0.05 two-sample test of proportions to detect a 15% absolute improvement in percentage of patients meeting the criteria with 544 patients (after adjusted for withdrawal and loss to follow-up); Test type: Superiority; p = 0.9238, Chi-squared, Corrected — Two-sided significance level = 0.05

2. Secondary Outcome: Calculated Cardiovascular (CVD) Risk Score at Two Years
Description: CVD risk score is obtained using the American Heart Association Risk Calculator (Goff et al, 2013). The calculator requires sex (all participants are male in this trial), age, race (White, African American, Other), HDL, total cholesterol, systolic blood pressure, diabetes (yes/no), treatment for hypertension (yes/no), smoker (yes/no), and provides a 10-year risk of atherosclerotic cardiovascular disease (ASCVD) events ranging from 0 (low risk) to 1 (high risk). The calculator documentation states that risk may be overestimated or underestimated for some subgroups of the race category "Other", therefore score is not calculated for any participants in this category.
Time Frame: Two years after completion of approximately 4-9 weeks of radiation therapy.
Population: Eligible participants with CVD risk score at two years.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Survivorship Care Plan) | Arm B (Enhanced Survivorship Care Plan)
Number analyzed (Participants) | 171 | 161
score on a scale | 0.257 (0.134) | 0.256 (0.135)
Statistical Analysis 1: Comparison: Arm A (Survivorship Care Plan) vs Arm B (Enhanced Survivorship Care Plan); Test type: Superiority; p = 0.5609, Mixed Models Analysis — Two-sided significance level = 0.05; Model included baseline CVD risk score, practice as random covariate (participants nested within practice) and treatment arm

3. Secondary Outcome: Components of the Primary Care Index (CPCI) Coordination of Care Subscale Score With Respect to the PCP (or Cardiologist if Patient Does Not Have a PCP)
Description: The Components of the Primary Care Index is a validated instrument specifically designed to measure aspects of primary care delivery from the patient's perspective. The coordination of care subscale measures the patients' perception of their physician's knowledge of other visits and visits to specialists, as well as the physician's follow-up of problems. Patients respond to six items, each on a 6-point Likert scale: strongly disagree (1), to strongly agree (6). The subscale score is the mean of the 6 items, with negatively-worded questions scored in reverse. A higher score indicates better coordination of care. All items had to be completed in order to calculate the score.
Time Frame: Two years after completion of approximately 4-9 weeks of radiation therapy.
Population: Eligible participants with two-year CPCI data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Survivorship Care Plan) | Arm B (Enhanced Survivorship Care Plan)
Number analyzed (Participants) | 204 | 193
score on a scale | 5.29 (0.96) | 5.46 (0.97)

4. Secondary Outcome: Patient Satisfaction With Care With Respect to the PCP (or Cardiologist if Patient Does Not Have a PCP)
Description: This 18-item instrument evaluates patient-reported outcomes related to satisfaction with cancer-related care. Patients respond to each item on a 5-point Likert scale from strongly disagree (1) to strongly agree (5). A total scale score is calculated by adding scores on all 18 items, ranging from 18 to 90. A higher score indicates higher satisfaction. All items had to be completed in order to calculate the score.
Time Frame: Two years after completion of approximately 4-9 weeks of radiation therapy.
Population: Eligible participants with two-year Patient Satisfaction with Care questionnaire data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Survivorship Care Plan) | Arm B (Enhanced Survivorship Care Plan)
Number analyzed (Participants) | 195 | 192
score on a scale | 81.96 (9.18) | 82.68 (11.80)

5. Other Pre Specified Outcome: Components of the Primary Care Index (CPCI) Coordination of Care Subscale Score With Respect to the Cancer Specialist
Description: as for outcome 3
Time Frame: Two years after completion of approximately 4-9 weeks of radiation therapy.
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Patient Satisfaction With Care With Respect to the Cancer Specialist
Description: as for outcome 4
Time Frame: Two years after completion of approximately 4-9 weeks of radiation therapy.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Arm A (SCP) | Arm B (Enhanced SCP)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT03860961/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/61/NCT03860961/ICF_001.pdf